CLINICAL TRIAL: NCT02948842
Title: Clostridium Histolyticum Collagenase Injection Treatment for Urethral Disease: a Prospective, Single-center, Open-label Study
Brief Title: Clostridium Histolyticum Collagenase Injection for Urethral Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHC
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Results first posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Urethral Stricture
MeSH Terms: conditions — Urethral Stricture | interventions — Microbial Collagenase; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): Patients will undergo instillation of local anesthesia (20 mL of 2% urethral lidocaine jelly), the patient will undergo cystoscopy, transurethral injection (via a 70 cm 4.8 Fr flexible cystoscopic needle with a 23 gauge needle tip manufactured by Laborie®, Ontario, Canada) of 0.08ml of XIAFLEX® (0.58 mg of XIAFLEX® mixed with 0.39 mL of sterile diluent) in a single location within the stricture, chased by an additional 0.25 mL of reconstituted XIAFLEX® to allow for clearance of the original 0.08 mL of reconstituted XIAFLEX® from the transurethral syringe into the urethral stricture.
  Interventions: Drug: Clostridium Histolyticum Collagenase; Other: Saline

INTERVENTIONS:
Drug: Clostridium Histolyticum Collagenase — 0.08ml of XIAFLEX® (0.58 mg of XIAFLEX® mixed with 0.39 mL of sterile diluent) in a single location within the stricture, chased by an additional 0.25 mL of reconstituted XIAFLEX® to allow for clearance of the original 0.08 mL of reconstituted XIAFLEX® from the transurethral syringe into the urethral stricture. This is based on 0.25 mL residual fluid that remains within the lumen of the injeTAK syringe. Thus, by adding the additional 0.25 mL of XIAFLEX® as a chase, we are expecting the original total of 0.08 mL of XIAFLEX® to be injected into the area of scarring.
  Other Names: XIAFLEX®
Other: Saline — 0.08ml of injectable normal saline
  Other Names: Injectable normal saline

SUMMARY:
The purpose of this study is to assess the efficacy of clostridium histolyticum collagenase (XIAFLEX®) in treating urethral strictures.

DETAILED DESCRIPTION:
This is an open-label, pilot study to explore the efficacy of clostridium histolyticum collagenase (XIAFLEX®) in treating urethral strictures. Subjects will be followed for 2 years from the initial drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age ≥ 18 years
* Failed prior proven conservative measures, including DVIU or balloon dilation of the stricture will be included in this study
* Able and willing to undergo regular intervention as well as evaluation as described below will be included in the study
* With a single stricture <2cm in size that can be identified on retrograde urethrogram or voiding cystourethrogram will be included in the study.
* Must agree not to participate in a clinical study involving another investigational drug or device throughout the duration of this study
* Must be competent to understand the information given in IRB approved ICF and must sign the form prior to the initiation of any study procedure

Exclusion Criteria:

* Has not yet undergone proven non-invasive measures, including DVIU or balloon dilation.
* Multiple strictures or a single stricture larger than 2cm in size, measured with retrograde urethrogram, voiding cystourethrogram, or urethral ultrasonography.
* Corporal spongiosum tissues < 5 mm in depth at proposed injection site
* Grade 5 spongiofibrosis
* Age <18
* Females
* Prior urethroplasty
* Urethral fistula
* History of penile cancer, prostate cancer, or urinary tract malignancy (bladder, urethral, ureteral, or kidney).
* History of radiation (external or brachytherapy) to the pelvic organs, penis or groin.
* History of autoimmune or inflammatory bowel disease
* Contraindication to suprapubic tube placement
* Pre-procedure PVR >250mL
* Allergy or sensitivity to CHC
* Bleeding disorder or anticoagulant use other than aspirin up to 150mg/day
* Untreated urinary tract infection
* Inability to perform intermittent self-catheterization
* Participation in another clinical study or treatment with an investigational drug or device
* Serious or active medical or psychiatric condition which, in the opinion of the Investigator, may interfere with treatment, assessment, or compliance with the protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas R Wiegand, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida - South Tampa Campus, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Santucci RA, Joyce GF, Wise M. Male urethral stricture disease. J Urol. 2007 May;177(5):1667-74. doi: 10.1016/j.juro.2007.01.041. PMID 17437780
- [Result] Chenoweth CE, Saint S. Urinary tract infections. Infect Dis Clin North Am. 2011 Mar;25(1):103-15. doi: 10.1016/j.idc.2010.11.005. Epub 2010 Dec 18. PMID 21315996
- [Result] Heyns CF, Steenkamp JW, De Kock ML, Whitaker P. Treatment of male urethral strictures: is repeated dilation or internal urethrotomy useful? J Urol. 1998 Aug;160(2):356-8. doi: 10.1016/s0022-5347(01)62894-5. PMID 9679876
- [Result] Hussain M, Greenwell TJ, Shah J, Mundy A. Long-term results of a self-expanding wallstent in the treatment of urethral stricture. BJU Int. 2004 Nov;94(7):1037-9. doi: 10.1111/j.1464-410X.2004.05100.x. PMID 15541123
- [Result] Zhang K, Qi E, Zhang Y, Sa Y, Fu Q. Efficacy and safety of local steroids for urethra strictures: a systematic review and meta-analysis. J Endourol. 2014 Aug;28(8):962-8. doi: 10.1089/end.2014.0090. Epub 2014 Jun 3. PMID 24745607
- [Result] Peak TC, Mitchell GC, Yafi FA, Hellstrom WJ. Role of collagenase clostridium histolyticum in Peyronie's disease. Biologics. 2015 Sep 29;9:107-16. doi: 10.2147/BTT.S65619. eCollection 2015. PMID 26491251
- [Result] Gelbard M, Goldstein I, Hellstrom WJ, McMahon CG, Smith T, Tursi J, Jones N, Kaufman GJ, Carson CC 3rd. Clinical efficacy, safety and tolerability of collagenase clostridium histolyticum for the treatment of peyronie disease in 2 large double-blind, randomized, placebo controlled phase 3 studies. J Urol. 2013 Jul;190(1):199-207. doi: 10.1016/j.juro.2013.01.087. Epub 2013 Jan 31. PMID 23376148
- [Result] Cavalcanti AG, Costa WS, Baskin LS, McAninch JA, Sampaio FJ. A morphometric analysis of bulbar urethral strictures. BJU Int. 2007 Aug;100(2):397-402. doi: 10.1111/j.1464-410X.2007.06904.x. PMID 17617144
- [Result] Sangkum P, Yafi FA, Kim H, Bouljihad M, Ranjan M, Datta A, Mandava SH, Sikka SC, Abdel-Mageed AB, Moparty K, Hellstrom WJ. Collagenase Clostridium histolyticum (Xiaflex) for the Treatment of Urethral Stricture Disease in a Rat Model of Urethral Fibrosis. Urology. 2015 Sep;86(3):647.e1-6. doi: 10.1016/j.urology.2015.06.013. Epub 2015 Jun 27. PMID 26126692

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 5
Completed | 1
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: 5 subjects enrolled in study, certain baseline data is available for only 4 subjects. One subject withdrew consent before all baseline visit procedures were completed.
Arm/Group | Treatment Group
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White: Hispanic | 1
  White: Non-Hispanic | 4
Height [Mean (Standard Deviation); unit: inches] | 70.8 (0.84)
Weight [Mean (Standard Deviation); unit: lbs] | 200 (19.0)
Stricture length [Mean (Standard Deviation); unit: cm] — The stricture length was determined via high-frequency ultrasound with lubricant instilled per urethra to delineate the urethral lumen and then measuring the maximum distance from normal diameter lumen to normal diameter lumen in a sagittal plane.
  cm | 0.96 (0.37)
Post void residual urine [Mean (Standard Deviation); unit: mL] — Post void residual urine (amount of urine that remains after urination) was measured via Laborie Portascan 3D ultrasound per standard clinical protocol immediately post-void. Population: One subject withdrew consent before all baseline procedures were completed, data not available for that subject
  mL
    number analyzed (Participants) | 4
    (all) | 64 (63)
Uroflowmetry [Mean (Standard Deviation); unit: mL/s] — Uroflowmetry was measured as the maximum flow rate as recorded via Laborie Urocap weight-based evaluation on a urine volume of at least 50mL as per standard clinical protocol. Population: One subject withdrew consent before all baseline procedures were completed, data not available for that subject
  mL/s
    number analyzed (Participants) | 4
    (all) | 8 (2.9)
Length of spongiofibrosis [Mean (Standard Deviation); unit: cm] — The length of spongiofibrosis was determine via high-frequency ultrasound with lubricant instilled per urethra to delineate the urethral lumen and then measuring the distance from normal-appearing spongiosal tissue to normal appearing tissue, traversing the structured segment, as determined by the investigator based on the echotexture. Population: One subject withdrew consent before all baseline procedures were completed, data not available for that subject
  cm
    number analyzed (Participants) | 4
    (all) | 0.51 (0.14)
Urethral stricture grade 2 [Count of Participants; unit: Participants] — Urethral stricture was graded based on ultrasound findings ranging from Grade 1 (short stricture with minimal spongiosal tissue involvement) to Grade 5 (full thickness/severe spongiosal involvement and at least 2 cm stricture length). Urethral stricture Grade 2 was short stricture with moderate spongiosal tissue involvement Population: One subject withdrew consent before all baseline procedures were completed, data not available for that subject
  Participants
    number analyzed (Participants) | 4
    (all) | 4
American Urological Association symptom score [Mean (Standard Deviation); unit: scores on a scale] — The American Urology Association questionnaire score is totaled based on 7 questions. Each question asks the subject to rate their symptom on a 5-point scale from "Not at All" (0) to "Almost Always" (5). The total score is based on adding rating marked for each question. The total runs from 0 to 35 points with higher scores indicating more severe symptoms.
  scores on a scale | 16 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Complication After Treatment
Description: Number of subjects with complication after treatment with clostridium histolyticum collagenase
Time Frame: 84 days
Population: Only 3 subjects were treated with study treatment. Two subjects withdrew prior to receiving study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Number of Patients Needing Further Intervention for Treatment of Urethral Stricture
Description: Further intervention - defined as any medical or surgical intervention for treatment of urethral stricture.
Time Frame: 2 years
Population: Only 3 subjects were treated with study treatment. Two subjects withdrew prior to receiving study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 3
Participants | 3

3. Secondary Outcome: Number of Subjects With Recurrence of Urethral Stricture
Description: Number of subjects with recurrence of urethral stricture
Time Frame: 2 years
Population: Only 3 subjects were treated with study treatment. Two subjects withdrew prior to receiving study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: Change From Baseline and 6 Weeks: American Urology Association Questionnaire Scores
Description: The American Urology Association questionnaire score is totaled based on 7 questions. Each question asks the subject to rate their symptom on a 5-point scale from "Not at All" (0) to "Almost Always" (5). The total score is based on adding rating marked for each question. The total runs from 0 to 35 points with higher scores indicating more severe symptoms.
Time Frame: 6 weeks
Population: Two subjects withdrew prior to receiving study treatment. Only 3 subjects were treated with study treatment. Only 2 out of 3 treated subjects completed 6 weeks follow-up.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 2
scores on a scale | -11.5 (3.5)

5. Secondary Outcome: Change From Baseline and 6 Months: American Urology Association Questionnaire Scores
Description: as for outcome 4
Time Frame: 6 months
Population: Two subjects withdrew prior to receiving study treatment. Only 3 subjects were treated with study treatment. Only 2 out of 3 treated subjects completed 6 months follow-up.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 2
scores on a scale | -2.5 (14.8)

6. Secondary Outcome: Change From Baseline and 9 Months: American Urology Association Questionnaire Scores
Description: as for outcome 4
Time Frame: 9 months
Population: Two subjects withdrew prior to receiving study treatment. Only 3 subjects were treated with study treatment. Only 1 out of 3 treated subjects completed 9 months follow-up.
Measure: Number; unit: scores on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 1
scores on a scale | -17

7. Secondary Outcome: Change From Baseline and 12 Months: American Urology Association Questionnaire Scores
Description: as for outcome 4
Time Frame: 12 months
Population: Two subjects withdrew prior to receiving study treatment. Only 3 subjects were treated with study treatment. Only 1 out of 3 treated subjects completed 12 months follow-up.
Measure: Number; unit: scores on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 1
scores on a scale | -19

8. Secondary Outcome: Change From Baseline and 2 Years: American Urology Association Questionnaire Scores
Description: as for outcome 4
Time Frame: 2 years
Population: Two subjects withdrew prior to receiving study treatment. Only 3 subjects were treated with study treatment. Only 1 out of 3 treated subjects completed 2 years follow-up.
Measure: Number; unit: scores on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 1
scores on a scale | -24

9. Secondary Outcome: Time to Urethral Stricture Recurrence
Time Frame: 2 years
Population: Only 3 subjects were treated with study treatment. Two subjects withdrew prior to receiving study treatment. None of the treated subjects had recurrence of urethral stricture.
Arm/Group | Treatment Group
Number analyzed (Participants) | 0

10. Secondary Outcome: Time to Additional Intervention for Urethral Stricture
Time Frame: 2 years
Population: Only 3 subjects were treated with study treatment. Two subjects withdrew prior to receiving study treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Treatment Group
Number analyzed (Participants) | 3
months | 6 [1 to 18]

11. Secondary Outcome: Change From Baseline and 6 Weeks: Obstructive Voiding Dysfunction (Uroflow)
Description: Obstructive voiding dysfunction defined as change in uroflow
Time Frame: 6 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Treatment Group
Number analyzed (Participants) | 2
mL/s | 1.5 (6.4)

12. Secondary Outcome: Change From Baseline and 6 Months: Obstructive Voiding Dysfunction (Uroflow)
Description: Obstructive voiding dysfunction defined as change in uroflow
Time Frame: 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Treatment Group
Number analyzed (Participants) | 2
mL/s | -5.5 (7.8)

13. Secondary Outcome: Change From Baseline and 9 Months: Obstructive Voiding Dysfunction (Uroflow)
Description: Obstructive voiding dysfunction defined as change in uroflow
Time Frame: 9 months
Population: as for outcome 6
Measure: Number; unit: mL/s
Arm/Group | Treatment Group
Number analyzed (Participants) | 1
mL/s | 3.6

14. Secondary Outcome: Change From Baseline and 12 Months: Obstructive Voiding Dysfunction (Uroflow)
Description: Obstructive voiding dysfunction defined as change in uroflow
Time Frame: 12 months
Population: as for outcome 7
Measure: Number; unit: mL/s
Arm/Group | Treatment Group
Number analyzed (Participants) | 1
mL/s | 5.8

15. Secondary Outcome: Change From Baseline and 18 Months: Obstructive Voiding Dysfunction (Uroflow)
Description: Obstructive voiding dysfunction defined as change in uroflow
Time Frame: 18 months
Population: Two subjects withdrew prior to receiving study treatment. Only 3 subjects were treated with study treatment. Only 1 out of 3 treated subjects completed 18 months follow-up.
Measure: Number; unit: mL/s
Arm/Group | Treatment Group
Number analyzed (Participants) | 1
mL/s | 19

16. Secondary Outcome: Change From Baseline and 2 Years: Obstructive Voiding Dysfunction (Uroflow)
Description: Obstructive voiding dysfunction defined as change in uroflow
Time Frame: 2 years
Population: as for outcome 8
Measure: Number; unit: mL/s
Arm/Group | Treatment Group
Number analyzed (Participants) | 1
mL/s | 9.2

17. Secondary Outcome: Change From Baseline and 6 Weeks: Obstructive Voiding Dysfunction (Post-void Residual Measurements)
Description: Obstructive voiding dysfunction defined as change in post-void residual measurements
Time Frame: 6 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Treatment Group
Number analyzed (Participants) | 2
mL | -41.5 (14.8)

18. Secondary Outcome: Change From Baseline and 6 Months: Obstructive Voiding Dysfunction (Post-void Residual Measurements)
Description: Obstructive voiding dysfunction defined as change in post-void residual measurements
Time Frame: 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Treatment Group
Number analyzed (Participants) | 2
mL | 175.5 (224.1)

19. Secondary Outcome: Change From Baseline and 9 Months: Obstructive Voiding Dysfunction (Post-void Residual Measurements)
Description: Obstructive voiding dysfunction defined as change in post-void residual measurements
Time Frame: 9 months
Population: as for outcome 6
Measure: Number; unit: mL
Arm/Group | Treatment Group
Number analyzed (Participants) | 1
mL | 125

20. Secondary Outcome: Change From Baseline and 12 Months: Obstructive Voiding Dysfunction (Post-void Residual Measurements)
Description: Obstructive voiding dysfunction defined as change in post-void residual measurements
Time Frame: 12 months
Population: as for outcome 7
Measure: Number; unit: mL
Arm/Group | Treatment Group
Number analyzed (Participants) | 1
mL | 46

21. Secondary Outcome: Change From Baseline and 18 Months: Obstructive Voiding Dysfunction (Post-void Residual Measurements)
Description: Obstructive voiding dysfunction defined as change in post-void residual measurements
Time Frame: 18 months
Population: as for outcome 15
Measure: Number; unit: mL
Arm/Group | Treatment Group
Number analyzed (Participants) | 1
mL | -48

22. Secondary Outcome: Change From Baseline and 2 Years: Obstructive Voiding Dysfunction (Post-void Residual Measurements)
Description: Obstructive voiding dysfunction defined as change in post-void residual measurements
Time Frame: 2 years
Population: as for outcome 8
Measure: Number; unit: mL
Arm/Group | Treatment Group
Number analyzed (Participants) | 1
mL | -15

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=3)
Dysuria (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 2
Worsening of urethral stricture (Renal and urinary disorders) | 2
Post void dribbling (Renal and urinary disorders) | 1 — Reported at 2 years follow-up
Right thigh pain (Renal and urinary disorders) | 1 — Following standard of care foley placement

LIMITATIONS AND CAVEATS:
These are first-in-human cases with collagenase clostridium histolyticum (CCH) treatment for urethral stricture, although number of treated patients is low. Future directions will hopefully include increased sample size through multi-institutional participation and adjunctive procedures designed to augment the proposed beneficial effects of CCH therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT02948842/Prot_SAP_000.pdf